CLINICAL TRIAL: NCT06138106
Title: Developing a Nutritional Supplement to Increase Collagen Synthesis in People
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 2110494
Record Dates: First submitted 2023-11-03; First posted 2023-11-18 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Dietary Supplements; Connective Tissue; Exercise
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Natural Product Supplement (Experimental): The participant will consume a dose of hydrolyzed collagen (20g) supplemented with vitamin C (100 mg), epicatechin (75 mg), vitamin E (350 iU) and stevia extract (225 mg).
  Interventions: Dietary Supplement: Natural Product Supplement
- Placebo (Placebo Comparator): The participant will consume a dose of hydrolyzed collagen (20g) supplemented with vitamin C (100 mg) and sweetener.
  Interventions: Dietary Supplement: Placebo control

INTERVENTIONS:
Dietary Supplement: Natural Product Supplement — Participants will have blood drawn before and one hour after consuming the natural product supplement. For 7-days the participants will perform load-bearing exercise and consume the supplement. On the final day, blood will be collected 4 hours after the final exercise bout.
  Arms: Natural Product Supplement
Dietary Supplement: Placebo control — Participants will have blood drawn before and one hour after consuming the placebo supplement. For 7-days the participants will perform load-bearing exercise and consume the supplement. On the final day, blood will be collected 4 hours after the final exercise bout.
  Arms: Placebo

SUMMARY:
The purpose of this study is to test whether a natural product supplement can potentiate the increase in collagen synthesis following the ingestion of collagen protein. The investigators have developed a model of natural (GRAS certified) products that stimulate collagen synthesis, in vitro. The investigators will determine whether the natural product supplement can potentiate the collagen synthetic response to the ingestion of collagen protein. Basal and fed serum will be isolated and these samples will be used to treat human engineered ligaments.

ELIGIBILITY:
Inclusion Criteria:

* Young healthy adults (18-30 y)

Exclusion Criteria:

* Pregnancy
* Smoking
* Receiving any medication that may interfere with the study outcomes

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-11-21 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Collagen protein synthesis | 7 days
  Collagen protein synthesis will be indirectly measured by measuring pro-collagen type I N-terminal propeptide (PINP) in the serum before and 4 hours after the last exercise bout (at day 7 of the protocol).

SECONDARY OUTCOMES:
Strength of ligament constructs | 60 minutes post-exercise
  Serum from participants will be used to treat engineered ligaments in order to measure the effect of the supplementation on the strength of the ligaments. The strength will be measured using the Instron bio puls 68SC-1 tension and compression machine.
Collagen content of ligament constructs | 60 minutes post-exercise
  Ligament constructs will be treated for 7 days with experimental feed medium containing serum obtained at baseline or post-prandial for determination of collagen content using a hydroxyproline assay.

CONTACTS AND LOCATIONS:
Overall Officials: Keith Baar, PhD, Principal Investigator — University of California, Davis
Locations (1):
- Hickey Laboratory, Davis, California, United States

IPD SHARING:
Plan to Share IPD: No